CLINICAL TRIAL: NCT04173767
Title: High-flow Nasal Cannula Oxygen Therapy for Ischemic Stroke Patients With Dysphagia and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHEN,CHUNG YAO, Physician, associate professor, department of physical medicine and rehabilitation, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG2H0011
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cerebral Infarction; Sleep Apnea, Obstructive; Deglutition Disorders
MeSH Terms: conditions — Cerebral Infarction; Sleep Apnea, Obstructive; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFNC (Experimental)
  Interventions: Device: high flow nasal cannula ventilation

INTERVENTIONS:
Device: high flow nasal cannula ventilation — High-flow nasal cannula (HFNC) ventilation therapy: supply heated & humidified air up to 60 L/min of flow; effects: positive end expiratory pressure effect, humidification.

SUMMARY:
High flow nasal cannula (HFNC) ventilation therapy was found to improve the severity of obstructive sleep apnea in non-stroke subjects. The investigators hypothesized that HFNC might be effective in stroke patients with dysphagia who needed nasogastric tube feeding and can not receive continuous positive airway pressure ventilation for obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke patients with dysphagia and obstructive sleep apnea who need nasogastric tube feedings

Exclusion Criteria:

* congestive heart failure, unconsciousness, chronic obstructive pulmonary disease, intracranial hemorrhage or malignancy, and unstable medical and neurological conditions
* central sleep apnea

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | once at polysomnography study night when receive high flow nasal cannula titration study
  respiratory inductance plethysmography sum (RIPsum) without calibration to score apnea and hypopnea events (American Academy of Sleep Medicine alternative criteria)
oxyhemoglobin desaturation index | once at polysomnography study night when receive high flow nasal cannula titration study
  number of times per hour of sleep that the blood's oxygen saturation level drops by ≥ 3% from baseline

SECONDARY OUTCOMES:
pulse wave velocity | baseline and 1 week after high flow nasal cannula therapy
  velocity (m/s) measured by SphygmoCor CPV system
heart rate variability | baseline and 1 week after high flow nasal cannula therapy
  measured by QHRV system (Medeia Ltd.)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Keelung, Taiwan